CLINICAL TRIAL: NCT04215445
Title: Effect of Sodium Glucose co Transporter 2 (SGLT2) Inhibition on Optical Coherence Tomography Angiography (OCT-A) Parameters in Diabetic Chronic Kidney Disease (CKD)
Brief Title: Effect of SGLT2 Inhibition on OCT-A Parameters in Diabetic CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Wan Haslina Wan Abdul Halim, Consultant Ophthalmologist-Cornea And Anterior Segment, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FF-2019-386
Record Dates: First submitted 2019-12-25; First posted 2020-01-02 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Diabetic Retinopathy; Chronic Kidney Diseases; Diabetes Mellitus
MeSH Terms: conditions — Diabetic Retinopathy; Renal Insufficiency, Chronic; Diabetes Mellitus | interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Proteinuric diabetic CKD (Active Comparator): Tab.empagliflozin 25mg once daily for 28 days
  Interventions: Drug: Empagliflozin 25 MG; Device: OCT-A
- Non-Proteinuric diabetic CKD (Active Comparator): Tab.empagliflozin 25mg once daily for 28 days
  Interventions: Drug: Empagliflozin 25 MG; Device: OCT-A

INTERVENTIONS:
Drug: Empagliflozin 25 MG — Tab.empagliflozin 25mg once daily for 28 days
  Other Names: Jardiance
Device: OCT-A — Optical coherence tomography angiography (OCT-A) is a non-invasive method to study the microvasculature of the retina and choroid.
  Other Names: Cirrus HD-OCT

SUMMARY:
Diabetes mellitus is a major and growing problem worldwide with many known micro and macrovascular complications. According to International Diabetes Federation, there were 285 million adults diagnosed with diabetes in 2010 and expected to increase to 439 million adult in 2030. It is a leading cause of chronic kidney disease (CKD) followed by hypertension, glomerulonephritis, and cystic kidney disease. Renal impairment patients metabolize and excrete drugs differently from patients with normal renal function and hence only limited number of oral hypoglycemic agent (OHA) available for them. One of the choices is sodium glucose co-transporter-2 inhibitor (SGLT2i) which is now widely used. Apart from its nephroprotective advantage, it also has additional benefit on cardiovascular and renal function based on EMPA-REG OUTCOME trial. One of the examples of SGLT2i is Empagliflozin (JARDIANCE) tablet, which has FDA U.S. Approval in 2014. It acts by reduces renal reabsorption of filtered glucose and lowers the renal threshold for glucose, thus increases urinary glucose excretion. It can cause osmotic diuresis, which may lead to intravascular volume contraction. Apart from its additional cardiovascular and nephroprotective effect, SGLT2 inhibitor might have additional protective effect to the eye. Nowadays, optical coherence tomography angiography (OCT-A) has emerged as one of a non-invasive methods to study the microvasculature of the retina and choroid. Many studies had discussed regarding-pre clinical changes present on OCT-A in patients without clinical diabetic retinopathy. These pre-clinical changes includes capillary dropout, microaneurysm, neovascularization, venous beading and enlargement of fovea avascular zone. However, there are minimal data and publications on different type of diabetic CKD with OCT-A parameters in diabetic patients. The purpose of this study is to determine the effect of short term SGLT2 inhibition on OCT-A parameters (fovea avascular zone (FAZ) size, vessel density and perfusion density) in diabetic CKD.

DETAILED DESCRIPTION:
This is a prospective, single-centred, open-labeled, randomized clinical trial conducted in ,University Kebangsaan Malaysia Medical Centre (UKMMC). This is also a Quasi-experimental study and all patients from Endocrine, Nephrology and Ophthalmology Clinic in UKM Medical Centre from November 2019 till November 2021 will be involved in this study. Patients who fulfill the inclusion criteria will be included in this study. All eligible subjects will be asked to sign an informed consent.

Participants will be randomized into two groups, diabetic patient with proteinuria and diabetic patient without proteinuria. Participants will be interviewed on demographic data (age, gender, race, blood pressure, Body Mass Index) will be taken. Urine sample and peripheral blood (2-3ml) is collected from patients in sterile container (EDTA tube) and will be sent for urine albumin creatinine ratio (ACR) and HbA1c test. The eye with best fundal and signal view on OCT-A will be chosen or if both eyes similar, right eye will be chosen. Pre-treatment tests fundus photo and OCT-A measurement will be taken at eye clinic after dilating the pupils with 1% tropicamide and 2.5% phenylephrine hydrochloride. Fundus examination is taken using a digital mydriatic retinal camera (Topcon Retinal Camera TRC-50DX (type 1A), Tokyo Japan. OCT-A measurement is taken by using Cirrus HD-OCT, 2016 Carl Zeiss Meditec.

Then Tab.empagliflozin 25mg once daily for 28 days will be given to both group of patients proteinuric and non proteinuric diabetic CKD. After 28 days, post-treatment tests of fundus examination and OCT-A measurement will be taken at eye clinic.

The statistical data analysis will be performed using statistical package for Social Science, version 22.0 (SPSS, Inc. Chicago III USA) for IOS. The OCT-A parameters studied (FAZ size, vessel density and perfusion density) will be used as main response variables. All variables will be defined by method of descriptive statistics. The analysis of quantitative variables includes a calculation of mean and standard deviation. T test will be performed to test the significant between the 2 groups. Correlation will be measured with Pearson correlation coefficient. A p <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Type 2 DM with CKD (eGFR 45 - 60 ml/min/1.7m2)
* Age between 35 and 65 year old
* Patients able to give informed consent to participate in the study.
* Patients previously not on tablet Empagliflozin

Exclusion Criteria:

* Heart or respiratory failure, recent MI, shock, hypotension
* Pregnancy or lactation.
* Known case of CKD due to other causes such as hypertension, renal calculi, analgesic nephropathy
* Patients with multiple diuretic use.
* Hypersensitivity reactions to SGLT2 group of agents
* Patient underwent previous ocular intervention (surgery, laser or intraocular injection) within 3 months
* Dense cataract which could obscured the fundal view and signal strength on OCT-A
* HbA1c more than 10%
* Systolic blood pressure more than 180mmHg

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Comparison of change in fovea avascular zone within retina of proteinuric and non-proteinuric chronic kidney disease patients treated with SGLT2-inhibitor | After 28 days of treatment
  Change in fovea vascular zone (FAZ) size (um2) from Baseline using Optical Coherence Tomography Angiography (OCT-A) post-SGLT-2 treatment
Comparison of change in retinal and choroidal vessel density in proteinuric and non-proteinuric chronic kidney disease patients treated with SGLT2-inhibitor | After 28 days of treatment
  Change in vessel density (mm-1) from Baseline using Optical Coherence Tomography Angiography (OCT-A) post-SGLT-2 treatment
Comparison of change in retinal and choroidal vascular perfusion density in proteinuric and non-proteinuric chronic kidney disease patients treated with SGLT2-inhibitor | After 28 days of treatment
  Change in perfusion density from Baseline using Optical Coherence Tomography Angiography (OCT-A) post-SGLT-2 treatment

CONTACTS AND LOCATIONS:
Overall Officials: Wan Haslina Wan Abdul Halim, M.D, Study Chair — Department of Ophthalmology, UKM Medical Centre
Locations (1):
- UKM Medical Centre, Kuala Lumpur, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] American Diabetes Association. 10. Microvascular Complications and Foot Care: Standards of Medical Care in Diabetes-2018. Diabetes Care. 2018 Jan;41(Suppl 1):S105-S118. doi: 10.2337/dc18-S010. PMID 29222381
- [Background] National Renal Registry Malaysia. 20th report of the Malaysian Dialysis & Transplant Registry 2013. Minist Heal Malaysia. 2013. Doi: 10.1143/JJAP.35.L657
- [Background] Port J Nephrol Hypert 2017; 31(2): 122-131 • Advance Access publication 29 May 2017. Diabetic Nephropathy and its two phenotypes: the proteinuric and non-proteinuric Regina Silva, Catarina Meng, Luís Coentrão
- [Background] Bolignano D, Zoccali C. Non-proteinuric rather than proteinuric renal diseases are the leading cause of end-stage kidney disease. Nephrol Dial Transplant. 2017 Apr 1;32(suppl_2):ii194-ii199. doi: 10.1093/ndt/gfw440. PMID 28340010
- [Background] Perez-Monteoliva, N. R., Robles et al. Non-proteinuric diabetic nephropathy is the main cause of chronic kidney disease. Journal of Hypertension: June 2018 - Volume 36 - Issue - p e11. doi: 10.1097/01.hjh.0000538992.55964.f1
- [Background] Garg AX, Kiberd BA, Clark WF, Haynes RB, Clase CM. Albuminuria and renal insufficiency prevalence guides population screening: results from the NHANES III. Kidney Int. 2002 Jun;61(6):2165-75. doi: 10.1046/j.1523-1755.2002.00356.x. PMID 12028457
- [Background] Rodriguez-Poncelas A, Garre-Olmo J, Franch-Nadal J, Diez-Espino J, Mundet-Tuduri X, Barrot-De la Puente J, Coll-de Tuero G; RedGDPS Study Group. Prevalence of chronic kidney disease in patients with type 2 diabetes in Spain: PERCEDIME2 study. BMC Nephrol. 2013 Feb 22;14:46. doi: 10.1186/1471-2369-14-46. PMID 23433046
- [Background] Penno G, Solini A, Bonora E, Fondelli C, Orsi E, Zerbini G, Trevisan R, Vedovato M, Gruden G, Cavalot F, Cignarelli M, Laviola L, Morano S, Nicolucci A, Pugliese G; Renal Insufficiency And Cardiovascular Events (RIACE) Study Group. Clinical significance of nonalbuminuric renal impairment in type 2 diabetes. J Hypertens. 2011 Sep;29(9):1802-9. doi: 10.1097/HJH.0b013e3283495cd6. PMID 21738053
- [Background] Retnakaran R, Cull CA, Thorne KI, Adler AI, Holman RR; UKPDS Study Group. Risk factors for renal dysfunction in type 2 diabetes: U.K. Prospective Diabetes Study 74. Diabetes. 2006 Jun;55(6):1832-9. doi: 10.2337/db05-1620. PMID 16731850
- [Background] Zinman B, Wanner C, Lachin JM, Fitchett D, Bluhmki E, Hantel S, Mattheus M, Devins T, Johansen OE, Woerle HJ, Broedl UC, Inzucchi SE; EMPA-REG OUTCOME Investigators. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015 Nov 26;373(22):2117-28. doi: 10.1056/NEJMoa1504720. Epub 2015 Sep 17. PMID 26378978
- [Background] Skrtic M, Cherney DZ. Sodium-glucose cotransporter-2 inhibition and the potential for renal protection in diabetic nephropathy. Curr Opin Nephrol Hypertens. 2015 Jan;24(1):96-103. doi: 10.1097/MNH.0000000000000084. PMID 25470017
- [Background] Komala MG, Panchapakesan U, Pollock C, Mather A. Sodium glucose cotransporter 2 and the diabetic kidney. Curr Opin Nephrol Hypertens. 2013 Jan;22(1):113-9. doi: 10.1097/MNH.0b013e32835a17ae. PMID 23042029
- [Background] JARDIANCE current prescribing information and medication guide, www.jardiance.com. Boerhringer Ingelheim International GambH.
- [Background] Vasilakou D, Karagiannis T, Athanasiadou E, Mainou M, Liakos A, Bekiari E, Sarigianni M, Matthews DR, Tsapas A. Sodium-glucose cotransporter 2 inhibitors for type 2 diabetes: a systematic review and meta-analysis. Ann Intern Med. 2013 Aug 20;159(4):262-74. doi: 10.7326/0003-4819-159-4-201308200-00007. PMID 24026259
- [Background] Nishimura R, Tanaka Y, Koiwai K, Inoue K, Hach T, Salsali A, Lund SS, Broedl UC. Effect of empagliflozin monotherapy on postprandial glucose and 24-hour glucose variability in Japanese patients with type 2 diabetes mellitus: a randomized, double-blind, placebo-controlled, 4-week study. Cardiovasc Diabetol. 2015 Jan 30;14:11. doi: 10.1186/s12933-014-0169-9. PMID 25633683
- [Background] Yoshizumi H, Ejima T, Nagao T, Wakisaka M. Recovery from Diabetic Macular Edema in a Diabetic Patient After Minimal Dose of a Sodium Glucose Co-Transporter 2 Inhibitor. Am J Case Rep. 2018 Apr 19;19:462-466. doi: 10.12659/ajcr.909708. PMID 29670074
- [Background] Mieno H, Yoneda K, Yamazaki M, Sakai R, Sotozono C, Fukui M. The Efficacy of Sodium-Glucose Cotransporter 2 (SGLT2) inhibitors for the treatment of chronic diabetic macular oedema in vitrectomised eyes: a retrospective study. BMJ Open Ophthalmol. 2018 Jul 23;3(1):e000130. doi: 10.1136/bmjophth-2017-000130. eCollection 2018. PMID 30123844
- [Background] SGLT2- inhibition with Empaglifozin Reduces Progression of Diabetic Retinopathy in Patients With High Risk of Diabetic Macular Edema (The SUPER-Trial)
- [Background] Thompson IA, Durrani AK, Patel S. Optical coherence tomography angiography characteristics in diabetic patients without clinical diabetic retinopathy. Eye (Lond). 2019 Apr;33(4):648-652. doi: 10.1038/s41433-018-0286-x. Epub 2018 Dec 3. PMID 30510234
- [Background] Goudot MM, Sikorav A, Semoun O, Miere A, Jung C, Courbebaisse B, Srour M, Freiha JG, Souied EH. Parafoveal OCT Angiography Features in Diabetic Patients without Clinical Diabetic Retinopathy: A Qualitative and Quantitative Analysis. J Ophthalmol. 2017;2017:8676091. doi: 10.1155/2017/8676091. Epub 2017 Jun 29. PMID 28761762
- [Background] Sandhu HS, Eladawi N, Elmogy M, Keynton R, Helmy O, Schaal S, El-Baz A. Automated diabetic retinopathy detection using optical coherence tomography angiography: a pilot study. Br J Ophthalmol. 2018 Nov;102(11):1564-1569. doi: 10.1136/bjophthalmol-2017-311489. Epub 2018 Jan 23. PMID 29363532
- [Background] Ashraf M, Nesper PL, Jampol LM, Yu F, Fawzi AA. Statistical Model of Optical Coherence Tomography Angiography Parameters That Correlate With Severity of Diabetic Retinopathy. Invest Ophthalmol Vis Sci. 2018 Aug 1;59(10):4292-4298. doi: 10.1167/iovs.18-24142. PMID 30167660
- [Background] Lee DH, Yi HC, Bae SH, Cho JH, Choi SW, Kim H. Risk factors for retinal microvascular impairment in type 2 diabetic patients without diabetic retinopathy. PLoS One. 2018 Aug 9;13(8):e0202103. doi: 10.1371/journal.pone.0202103. eCollection 2018. PMID 30092018
- [Background] Ting DSW, Tan GSW, Agrawal R, Yanagi Y, Sie NM, Wong CW, San Yeo IY, Lee SY, Cheung CMG, Wong TY. Optical Coherence Tomographic Angiography in Type 2 Diabetes and Diabetic Retinopathy. JAMA Ophthalmol. 2017 Apr 1;135(4):306-312. doi: 10.1001/jamaophthalmol.2016.5877. PMID 28208170
- [Background] Cheung CY, Tang F, Ng DS, Wong R, Lok J, Sun Z, Tso T, Lam A, Brelen M, Chong KK, Luk AO, Chan JC, Wong TY, Tham CC. The Relationship of Quantitative Retinal Capillary Network to Kidney Function in Type 2 Diabetes. Am J Kidney Dis. 2018 Jun;71(6):916-918. doi: 10.1053/j.ajkd.2017.12.010. Epub 2018 Feb 28. No abstract available. PMID 29501263
- [Background] CIRRUS HD-OCT User Manual- Models 500, 5000 ©2016 Carl Zeiss Meditec, Inc